CLINICAL TRIAL: NCT01091155
Title: COMPRES - COMpression Anastomosis Ring (CAR™ 27/ColonRing™) Post maRketing Evaluation Study
Acronym: COMPRES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: novoGI (Industry)
Collaborators: Atlanta Colon & Rectal Surgery, Atlanta, GA (Other); FPMG Center for Colon & Rectal Surgery (Unknown); Lester E. Cox Medical Centers (Other); UCI Medical Center Irvine CA (Unknown); Endeavor Health (Other); St.Louis University hospital MO (Unknown); University of Southern California (Other); Bnai Zion Medical Center (Other Government); Barmherzig Brueder (Unknown); Catharina Ziekenhuis Eindhoven (Other); Ziekenhuis Oost-Limburg (Other); University Hospital, Gasthuisberg (Other); Klinikum Neuperlach (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Protocol COMPRES 23/11/2009; NCT00859924 (obsolete NCT alias)
Record Dates: First submitted 2010-03-19; First posted 2010-03-23 (Estimated); Results first posted 2013-10-25 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-08

CONDITIONS: Colorectal Surgery
Keywords: Colon Anastomosis; Rectum Anastomosis; Intestine; Colorectal Surgery; Colorectal Anastomosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ColonRing TM (Experimental)
  Interventions: Device: ColonRing (Colorectal anastomosis)

INTERVENTIONS:
Device: ColonRing (Colorectal anastomosis) — Creation of a colorectal compression anastomosis

SUMMARY:
The performance of the ColonRing™ will be comparable to or better than the reported performance of staplers.

DETAILED DESCRIPTION:
The proposed study is a post marketing study intended to gather and record additional data to further evaluate the performance of the ColonRing™ device in regards to the creation of a colorectal anastomosis.

The study objective is to evaluate the performance of the ColonRing™ in the creation of a circular anastomosis in colorectal procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years old.
2. BMI < 34.
3. Subject is planned to undergo a non-emergency (i.e., elective) operation with the creation of an anastomosis using the ColonRing™.
4. Subject signs and dates a written informed consent form (ICF) and indicates an understanding of the study procedures.

Exclusion Criteria:

1. Subject has a known allergy to nickel.
2. Subject is planned to undergo an emergency procedure or has a diagnosis of bowel strangulation, peritonitis, bowel perforation, local or systemic infection, ischemic bowel,carcinomatosis.
3. Subject has participated in another clinical study which may affect this study's outcomes within the last 30 days.
4. Subject's ASA (American Society of Anesthesiology) score 4 or 5.
5. Subject has a concurrent or previous invasive pelvic malignancy.
6. Subject has a systemic or incapacitating disease.
7. Subject has extensive local disease in the pelvis.
8. Subject requires more than one anastomosis during the surgery.
9. Women who are known to be pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2010-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eran Choman, Msc, Study Director — novoGI
Locations (13):
- United States (7):
  - UCI Medical Center, Irvine, California
  - University of Southern California Health Sciences Campus, Los Angeles, California
  - FPMG Center for Colon & Rectal Surgery, Orlando, Florida
  - Southern Regional Medical Center, Riverdale, Georgia
  - NorthShore University Health System, Evanston, Illinois
  - Lester E. Cox Medical Center, Springfield, Missouri
  - St. Louis University Hospital, St Louis, Missouri
- KH Barmherzig Brueder, Vienna, Austria
- Belgium (2):
  - Ziekenhuis Oost Limburg, Genk
  - University Hospital Gasthuisberg, Leuven
- Klinikum Neuperlach, Munich, Germany
- Bnai Zion Medical Center, Haifa, Israel
- Catharina Ziekenhuis, Eindhoven, Netherlands

REFERENCES:
- See also: Click here for more information about study device (sponsor's web site) — http://www.nitisurgical.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- ColonRing TM: ColonRing (Colorectal anastomosis) : Creation of a colorectal compression anastomosis
Period: Overall Study
Arm/Group | ColonRing TM
Started | 288
Completed | 279
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | ColonRing TM
Number analyzed (Participants) | 288
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 177
  >=65 years | 111
Age Continuous [Mean (Standard Deviation); unit: years] | 60 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146
  Male | 142
Region of Enrollment [Number; unit: participants]
  United States | 127
  Belgium | 83
  Austria | 46
  Israel | 13
  Germany | 9
  Netherlands | 10

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate Rate of Anastomotic Leaks Related to the Use of the ColonRing™ Device, at 1 Month
Description: Anastomotic leakage will be defined as clinical symptoms such as fever or sepsis in combination with pelvic abscess, rectovaginal fistula or peritonitis within 30 days postoperatively leading to a clinical and / or radiological interventional procedure of the subject, or operation that confirms the leakage which has been determined to be related to the device.
Time Frame: Approx. 1 year
Reporting Status: Not Posted

2. Secondary Outcome: Rate of Other Device Related Complications and Other Parameters During Hospitalization and Post Procedure.
Description: The post operative parameters that will be measured during hospitalization period:
  1. Hospitalization time (two dates will be recorded: ready for discharge and discharge). The later noting where the subject was discharged to - e.g. nursing home or home
  2. First day to first postoperative flatus
  3. First day to first postoperative bowel movements
  4. First day of first postoperative toleration of liquids and solids (time to "keeping them down")
Time Frame: 30 days post op
Reporting Status: Not Posted

3. Primary Outcome: Device Related Leak Rate up to 30 Days Post op
Description: as for outcome 1
Time Frame: 30 days post op
Measure: Number; unit: participants
Arm/Group | ColonRing TM
Number analyzed (Participants) | 279
participants | 4

ADVERSE EVENTS:
Arm/Group | ColonRing TM
Serious Adverse Events (participants affected / at risk) | 26/279
Other Adverse Events (participants affected / at risk) | 0/279
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ColonRing TM (N=279)
Leak (Surgical and medical procedures) | 16 (26)
Abscess (Surgical and medical procedures) | 8 (26)
Fistula (Surgical and medical procedures) | 2 (26)

LIMITATIONS AND CAVEATS:
The study had acceptable rate of AE, and technical problems.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
14.1 Review. Institution may publish the results of the Study, based on information collected or generated by Institution and Principal Investigator within the framework thereof, subject to the provisions of this section. In any event, however, no publication, presentation in any forum or any other form of disclosure with respect to the Study or the results thereof will be made prior to the publication of the Joint Publication without Sponsor's prior written consent.